CLINICAL TRIAL: NCT02353130
Title: Development Of Cortical Metrics Assessment Outcome Measures in Response to Memantine Treatment in Autism Spectrum Disorders
Brief Title: Cortical Metrics Assessment Outcome Measure Development in Autism With Memantine Treatment
Status: Withdrawn | Type: Observational
Why Stopped: Protocol did not continue once Investigator relocated to another institution
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1996
Record Dates: First submitted 2015-01-27; First posted 2015-02-02 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2015-10

CONDITIONS: Autism Spectrum Disorders
Keywords: autism spectrum disorders; memantine; cortical metrics; sensory testing
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Memantine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Memantine-XR: Boys ages 8-12 with ASD treated with Memantine-XR daily for 8 weeks
  Interventions: Drug: Memantine-XR

INTERVENTIONS:
Drug: Memantine-XR — Participants will begin with 7mg Memantine XR® daily for a minimum of one week before increasing to an optimal dose of 14 mg daily. It is suggested that participants be titrated to the optimal dose by week 2 so that they may remain on 14mg for at least 6 weeks. Morning dosing is suggested, but can be flexible.
  Other Names: Namenda-XR

SUMMARY:
Specific Aim 1: Obtain proof of concept evidence that cortical metrics will change in response to treatment with Memantine extended release (XR)®, an agent that modulates n-methyl d-asptartate (NMDA) receptor activation, in children with autism spectrum disorders (ASD) who clinically demonstrate treatment response.

Hypothesis1: Children with ASD who have dramatic clinical response to Memantine XR® will exhibit changes in their cortical metrics, which will differ less from neurotypical children. Subjective ratings of improvement will be correlated with the change in cortical metrics.

The completion of these aims will be essential to design a larger federally funded trial to validate cortical metrics as an outcome measure in a more heterogeneous pediatric ASD sample. Specifically, the feasibility data obtained may demonstrate the potential for detecting changes in cortical metrics over time, so that a larger grant could focus on determining how sensitive and clinically relevant changes in cortical metrics are or may indicate the need to explore different interventions to use in a validation study. We have chosen to use Memantine XR® because of its impact on NMDA neurotransmission, its current evaluation in a large multi-site randomized ASD clinical trial whose initial results are expected shortly, and our own observations of clinical improvements and good tolerability in the ongoing trial.

DETAILED DESCRIPTION:
Youth with ASD ages 8-12 years will undergo cortical metrics testing (testing of ability to discriminate the vibration of small brushes on the tops of the hand under various conditions) prior to treatment with memantine XR. They will then be treated with memantine XR target dose of 14milligrams daily for 8 weeks. At the end of 8 weeks, cortical metrics testing will be repeated. Within-subject changes in the cortical metrics testing between baseline and endpoint will be examined and described. Potential relationships between changes in clinical rating scales and cortical metrics will be examined. Data will be utilized to inform a decision about continuing to explore the utility of cortical metrics to detect changes in brain function in youth with ASD in response to therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male Boys ages 8-12 with ASD (confirmed with ADOS-2 and DSM-5 checklist at screening)
* IQ's should be within the normal range (≥ 70) (by prior testing or Stanford-Binet 5 at screening)
* Primary caretaker is able to participate in study appointments as is clinically indicated.
* Ability of child to participate in all aspects of the protocol per investigator clinical judgment

Exclusion Criteria:

* No new educational or behavioral intervention within 4 weeks of baseline.
* No history of non-febrile seizures, other neurological disorders, or comorbid psychiatric disorders.
* Impairment of renal function
* Evidence or history of malignancy
* Any significant medical conditions including but not limited to hematological, endocrine, respiratory, hepatic, cardiovascular or gastrointestinal disease
* Patients who, in the investigator's opinion, might not be suitable for the study
* Significant risk of suicidality based on investigator judgment
* History of hypersensitivity reaction to Memantine, dextromethorphan, amantadine or any other NMDA antagonists
* Changes in psychotropic medications within 4 weeks of baseline visit

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: 15 boys with ASD (8-12 years old) will receive Memantine XR®.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
cortical metrics (a mathematical plot of tactile responsivity in 3 dimensions) | 8 weeks
  a mathematical plot of tactile responsivity in 3 dimensions

SECONDARY OUTCOMES:
Clinical Global Impressions - Improvement Score. | 8 weeks
  ratings of 1 or 2 indicate clinically meaningful response
PDD-BI SV change 0-8 | 8 weeks
  18 item caregiver completed questionnaire about social functioning
ABC-SW subscale score 0-8 | 8 weeks
  13 item caregiver completed questionnaire about social problems

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- [Derived] Brignell A, Marraffa C, Williams K, May T. Memantine for autism spectrum disorder. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013845. doi: 10.1002/14651858.CD013845.pub2. PMID 36006807